CLINICAL TRIAL: NCT00124683
Title: Optimizing Treatment for Schizophrenic Smokers
Brief Title: Treating Nicotine Dependence in Schizophrenic Individuals: Effectiveness of Bupropion - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-13672-1; R01-13672-1; DPMC
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2007-08

CONDITIONS: Tobacco Use Cessation; Tobacco Use Disorder; Schizophrenia
Keywords: nicotine dependence
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use Disorder; Schizophrenia | interventions — Bupropion; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Nicotine Patch + Bupropion
  Interventions: Drug: Bupropion; Drug: nicotine transdermal patch
- 2 (Placebo Comparator): Nicotine patch + placebo
  Interventions: Drug: nicotine transdermal patch

INTERVENTIONS:
Drug: Bupropion
  Arms: 1
Drug: nicotine transdermal patch

SUMMARY:
Schizophrenic individuals are typically nicotine dependent smokers who find it difficult to quit smoking. The purpose of this study is to determine the effectiveness of bupropion SR (commonly known as Zyban) in combination with a nicotine transdermal patch (NTP), in helping schizophrenic individuals quit smoking. In addition, this study will evaluate how the combination of bupropion SR and NTP affects psychiatric symptoms and medication side effects.

DETAILED DESCRIPTION:
Past research on the use of the NTP, atypical antipsychotics, and bupropion in schizophrenic individuals to aid in smoking cessation has been encouraging. The purpose of this study is to compare bupropion SR to a placebo to determine its effectiveness when used in combination with an NTP to help schizophrenic individuals quit smoking.

Participants in this double-blind, placebo-controlled study will be randomly assigned to receive either the NTP (21 mg/day) and placebo or the NTP and bupropion SR (300 mg/day). Participants will begin taking one pill each day of bupropion SR (150 mg/day) or placebo at the start of the second week of the study. After three days, the dose of bupropion SR or placebo will increase to 2 pills each day. Participants will continue this dosing regimen until the end of Week 10. Throughout the 10-week study, participants will receive weekly group therapy.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder and nicotine dependence
* Fagerstrom Test for Nicotine Dependence (FTND) score greater than 5
* Smokes at least 20 cigarettes per day (1 pack per day)
* Expired breath CO level > 10 ppm and cotinine level > 210 ng/ml at the baseline measurement
* Currently taking a stable dose of antipsychotic
* Complete remission from positive symptoms of psychosis as judged by a psychiatric evaluation

Exclusion Criteria:

* Meets criteria for current abuse or dependence for any alcohol or illicit substance within the past month
* History of hypersensitivity to bupropion or the nicotine transdermal patch (NTP)
* Current diagnosis of a serious documented medical disorder that would make bupropion treatment risky OR results of psychiatric/medical screening that suggest a reason for concern (e.g., a history of severe heart, liver, or kidney disease or diabetes mellitus)
* Currently taking monoamine oxidase inhibitors or bupropion (Zyban or Wellbutrin)
* Currently taking diabetes mellitus medications, St. John's Wort, appetite suppressants, ephedrine-containing medications, theophylline, clonidine, reserpine, methyldopa, or anti-anginal medications (e.g., beta-blockers, calcium channel blockers, nitroglycerin preparations)
* History of schizoaffective disorder and not stabilized on a mood stabilizer (e.g., lithium, valproate, carbamazepine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2001-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
7 day point prevalence of cigarette abstinence | End of trial (week 10)

SECONDARY OUTCOMES:
Craving | assessed weekly
Medication compliance | assessed weekly
Depression | assessed at weeks 1, 4, 7, 10 and at six-month followup
Withdrawal symptoms | assessed weekly and at six month followup
Schizophrenic symptoms | assessed at weeks 1, 4, 7, 10 and at six-month followup

CONTACTS AND LOCATIONS:
Overall Officials: Tony P George, M.D., Principal Investigator — Yale University

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] George TP, Vessicchio JC, Sacco KA, Weinberger AH, Dudas MM, Allen TM, Creeden CL, Potenza MN, Feingold A, Jatlow PI. A placebo-controlled trial of bupropion combined with nicotine patch for smoking cessation in schizophrenia. Biol Psychiatry. 2008 Jun 1;63(11):1092-6. doi: 10.1016/j.biopsych.2007.11.002. Epub 2007 Dec 21. PMID 18096137